CLINICAL TRIAL: NCT06687551
Title: JAK Inhibitor Dose TAPering Strategy Study in Low Disease Activity Rheumatoid Arthritis Patients
Brief Title: JAK Inhibitor Dose TAPering Strategy Study
Acronym: JAK-TAP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/23/0373; 2023-509788-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-29; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Rhumatoid Arthisis
Keywords: JAK-inhibitor; dose reduction; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib; GLPG0634; tofacitinib; upadacitinib

STUDY DESIGN:
Intervention Model Description: This study will take the format of a prospective therapeutic research. The design will be a pragmatic multicentre open-label simple-blinded, non-inferiority randomised controlled trial with two parallel groups, ratio 1:1, comparing the two following groups:
  1. JAK inhibitor dose-tapering strategy.
  2. JAK inhibitor continuous therapy strategy.
Who Masked: Investigator
Masking Description: This study will be a simple blinded trial, because the investigator in charge of the primary outcome assessment (CDAI) will be blinded to the randomisation arm. This independent investigator will also collect all the disease activity index (CDAI, SDAI and DAS28-ESR) in the other follow-up visits, since the results of the definition of the flares and strategy changes will be based on these disease activity index.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JAK inhibitor dose-tapering strategy (Experimental): The dose-tapering strategy will depend on the JAK inhibitor taken by the patient. It will be based on a 50% dose-reduction every 6 months and will comprise 2 steps:
  A. Treatment with baricitinib 4 mg daily:
  * Step 1 (after randomization): baricitinib 2mg daily.
  * Step 2 (in case of CDAI ≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): baricitinib 2mg every other day.
  B. Treatment with filgotinib 200 mg daily:
  * Step 1 (after randomisation): filgotinib 100 mg daily.
  * Step 2 (in case of CDAI ≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): filgotinib 100mg every other day.
  C. Treatment with tofacitinib 5 mg twice daily or tofacitinib 11mg daily:
  * Step 1 (after randomisation): tofacitinib 5 mg once daily.
  * Step 2 (in case of CDAI ≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): tofacitinib 5 mg every other day.
  D. Treatment with upadacitinib 15 mg daily:
  • Step 1 (after randomisat
  Interventions: Drug: Baricitinib (LY3009104) 4 mg; Drug: filgotinib 200mg/day; Drug: Tofacitinib 5 mg twice daily; Drug: Upadacitinib 15 MG
- JAK inhibitor continuous therapy strategy (Active Comparator): Full dose will be considered in patient taking:
  * Baricitinib 4mg/day
  * Filgotinib: 200mg/day
  * Tofacitinib : 5mg twice daily or 11mg/day
  * Upadacitinib: 15mg/day
  Interventions: Drug: Baricitinib (LY3009104) 4 mg; Drug: filgotinib 200mg/day; Drug: Tofacitinib 5 mg twice daily; Drug: Upadacitinib 15 MG

INTERVENTIONS:
Drug: Baricitinib (LY3009104) 4 mg — Treatment with baricitinib 4 mg daily
  * Step 1 (after randomization): baricitinib 2mg daily
  * Step 2 (in case of CDAI≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): baricitinib 2mg every other day
  Arms: JAK inhibitor dose-tapering strategy
Drug: filgotinib 200mg/day — Treatment with filgotinib 200 mg daily
  * Step 1 (after randomisation): filgotinib 100 mg daily
  * Step 2 (in case of CDAI≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): filgotinib 100mg every other day
  Arms: JAK inhibitor dose-tapering strategy
Drug: Tofacitinib 5 mg twice daily — Treatment with tofacitinib 5 mg twice daily or tofacitinib 11mg daily
  * Step 1 (after randomisation): tofacitinib 5 mg once daily
  * Step 2 (in case of CDAI≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): tofacitinib 5 mg every other day
  Arms: JAK inhibitor dose-tapering strategy
Drug: Upadacitinib 15 MG — Treatment with upadacitinib 15 mg daily
  * Step 1 (after randomisation): upadacitinib 15 mg every other day
  * Step 2 (in case of CDAI≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): upadacitinib 15 mg every 4 days
  Arms: JAK inhibitor dose-tapering strategy
Drug: Baricitinib (LY3009104) 4 mg — use of JAK inhibitor at full dose until the end of the protocol
  Arms: JAK inhibitor continuous therapy strategy
Drug: filgotinib 200mg/day — use of JAK inhibitor at full dose until the end of the protocol
  Arms: JAK inhibitor continuous therapy strategy
Drug: Tofacitinib 5 mg twice daily — use of JAK inhibitor at full dose until the end of the protocol
  Arms: JAK inhibitor continuous therapy strategy
Drug: Upadacitinib 15 MG — use of JAK inhibitor at full dose until the end of the protocol
  Arms: JAK inhibitor continuous therapy strategy

SUMMARY:
This study aims to assess the feasibility of tapering JAK inhibitors in rheumatoid arthritis patients in low disease activity by comparing a group of patients tapering the JAK inhibitor dosage to a group of patients continuing the full-dose.

Participants will:

* Either take

  1. JAK inhibitor dose-tapering strategy.
  2. JAK inhibitor continuous therapy strategy.
* Visit the clinic once every 3 months for checkups and tests
* Keep a diary of their treatment intake and symptoms

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an autoimmune disease leading to inflammation of the synovium and joint erosions, responsible for joint damage leading to pain, functional impairment, work loss and disability. The prognosis of the disease has been greatly improved for 20 years with the use of Disease-Modifying Anti-Rheumatic Drugs (DMARDs) and especially biologic DMARDs.

It is recommended to target remission when initiating a DMARD and to assess patients according to a treat-to-target approach in order to adapt therapy. Once sustained remission is achieved, a decrease in the targeted therapeutic DMARD dose should be considered, according to the recommendations, in order to reduce the risk of adverse events and medical costs. Indeed, targeted DMARDs have considerably increased medical costs linked to RA and studies assessing medical economic impact of bDMARD down-titration on medical costs highlighted the cost-utility of such strategies.

JAK inhibitors, a novel class of targeted therapies have proved to be very effective in treating inflammation and preventing structural progression in RA. However, awareness has recently been raised regarding the safety of JAK inhibitor in the treatment of RA, with particular emphasis on tofacitinib. Indeed, tofacitinib seems to increase the risk of thromboembolism events, infections, neoplasia and major cardiovascular events in comparison to anti-TNF in RA, with a dose-effect.

To date, we have very little data regarding the feasibility of a JAK inhibitor dose-tapering strategy. As a dose-related effect was apparent in terms of major adverse events, we assume that JAK inhibitor dose-tapering strategy might reduce the risk of serious adverse events, without increasing the risk of major flares and thus be beneficial for the patient.

The aim of the study will be to compare a dose-tapering strategy versus therapy continuation in rheumatoid arthritis patients in low disease activity treated with JAK inhibitors on the risk of losing low disease activity despite rescue therapy at 12 months.

1) The dose-tapering strategy will depend on the JAK inhibitor taken by the patient. It will be based on a 50% dose-reduction every 6 months and will comprise 2 steps:

A. Treatment with baricitinib 4 mg daily:

* Step 1 (after randomization): baricitinib 2mg daily.
* Step 2 (in case of CDAI ≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): baricitinib 2mg every other day.

B. Treatment with filgotinib 200 mg daily:

* Step 1 (after randomisation): filgotinib 100 mg daily.
* Step 2 (in case of CDAI ≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): filgotinib 100mg every other day.

C. Treatment with tofacitinib 5 mg twice daily or tofacitinib 11mg daily:

* Step 1 (after randomisation): tofacitinib 5 mg once daily.
* Step 2 (in case of CDAI ≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): tofacitinib 5 mg every other day.

D. Treatment with upadacitinib 15 mg daily:

* Step 1 (after randomisation): upadacitinib 15 mg every other day.
* Step 2 (in case of CDAI ≤ 10 AND CRP level below the laboratory standard; 6 months after starting step1): upadacitinib 15 mg every 4 days.

Management of flares:

1. In case of flare, diagnosed during a scheduled visit: the management of the flare will be standardized by a rescue therapy including a glucocorticoid course and returning to the previous step of JAK inhibitor dose. If the flare is not resolved after the rescue therapy, the patient will be considered in failure of the strategy.
2. In case of flare between two scheduled visits, an additional visit will be scheduled by the clinical center to confirm the flare by the physician. If the flare is confirmed, the patient will have the standardized flare management as described above.

2) Patients randomised to the control group will have to continue the JAK inhibitor at full dose until the end of the protocol:

* In case of baricitinib: baricitinib 4mg/day.
* In case of filgotinib: filgotinib 200mg/day.
* In case of tofacitinib: tofacitinib 5mg twice daily or 11mg/day.
* In case of upadacitinib: upadacitinib 15mg/day.

Management of flares:

1. In case of flare, diagnosed during a scheduled visit: the management of the flare will be standardized by a rescue therapy with a glucocorticoid course. If the flare is not resolved after the rescue therapy, the patient will be considered in failure of the strategy.
2. In case of flare between two scheduled visits, an additional visit will be scheduled by the clinical center to confirm the flare by the physician. If the flare is confirmed, the patient will have the standardized flare management as described above.

Patients with co-medication with sDMARD or glucocorticoids < 5mg/d will have to keep a stable dose of their treatment during the 12 months of the study in both groups.

ELIGIBILITY:
The inclusion criteria will be

1. Aged ≥ 18 years at baseline.
2. Rheumatoid arthritis defined by the ACR/EULAR criteria.
3. Treated with a JAK inhibitor, full dose for at least 6 months.
4. The JAK inhibitor is prescribed as monotherapy or combined with a csDMARD with a stable dosage for at least 3 months before inclusion.
5. Being in LDA (CDAI≤10) for at least 6 months.
6. With a CRP level below the laboratory standard within the month before the inclusion visit.
7. Women of childbearing potential (WCBP) must have a negative pregnancy test before starting study

The non-inclusion criteria will be:

1. Concomitant disease needing to be treated by the JAK inhibitor at full-dose (for example inflammatory bowel disease).
2. Patient with a history of JAK-inhibitor dose reduction/spacing before enrollment in the study with the JAK-inhibitor currently being taken.
3. Evidence of flare-up within the last 6 months prior to the inclusion.
4. Patient who received glucocorticoids > 5mg/day in the 3 months prior the inclusion because of the disease activity of the RA.
5. Patient requiring corticoid joint injections in the 3 months prior to inclusion or with scheduled joint injections, to control disease activity.
6. Patient at risk for complication according to the ANSM (60) (current or past smokers, patients at risk of VTE, cancer or major cardiovascular problems, aged ≥ 65 years) at baseline AND currently taking baricitinib or filgotinib.
7. Patient taking associated bDMARD (including anti-TNF, anti-IL6, anti-CD20, abatacept, anti-IL17, anti-IL12/23, anti-IL23, anti-IL1, anti-BAFF, anti-IL5 pathways).
8. Patient taking immunotherapy for neoplasia.
9. Surgery scheduled in the next 12 months.
10. Fibromyalgia according to the physician's opinion.
11. Anticipated poor compliance with the strategy.
12. Patient with any condition that would prevent participation in the study and completion of the study procedures, including language limitation.
13. Alcohol and/or drug misuse as determined by the investigator.
14. Pregnancy or breastfeeding.
15. Non-affiliation to the French Social Security System.
16. Patient unwilling to sign the informed consent form.
17. Patient under legal protection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
proportion of patients still receiving a JAK-inhibitor | 12 post baseline
  The primary outcome of this study will be the proportion of patients still receiving a JAK-inhibitor and being in CDAI low disease activity at 12 months.
  The size of the effect will be given in the form of the difference in proportion between the two treatment groups with a two-sided confidence interval at 95%. Non-inferiority will be assessed with this interval. Non-inferiority will be concluded if the lower limit of the 95% confidence interval does not exceed the non-inferiority margin of 10% of the difference in proportion.

SECONDARY OUTCOMES:
Flare occurence | first flare post baseline
  The delay between the inclusion visit and the first flare diagnosed by a physician.
  Two definitions of flare can be used for this criterion:
  * A flare defined by a CDAI > 10 at any visit.
  * A major flare at any visit, based on the OMERACT definition which is:
    * An increase in the DAS28-ESR score of more than 1.2 compared to baseline score,
    * OR a DAS28-ESR score increase of more than 0.6 compared to the baseline score AND the current DAS28-ESR score being above 3.2.